CLINICAL TRIAL: NCT06701968
Title: A Healthy Nordic Diet to Reduce the Progression of Atherosclerosis in Individuals with Coronary Heart Disease: a Secondary Prevention Trial
Brief Title: Effects of a Healthy Nordic Diet on Atherosclerosis in Patients with Coronary Heart Disease
Acronym: NORDHEART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: Falu Hospital (Other)
Responsible Party: Principal Investigator, Ulf Risérus, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NORDHEART trial
Record Dates: First submitted 2024-11-19; First posted 2024-11-22 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-11

CONDITIONS: Coronary Disease; Coronary Arteriosclerosis; Myocardial Infarction; Chronic Coronary Syndrome; MASLD; Type 2 Diabetes
Keywords: Diet; Secondary prevention; Coronary plaque regression; Atherosclerosis; Type 2 diabetes; Coronary heart disease; Myocardial infarction; Coronary computed tomography angiography; Healthy nordic diet; NAFLD
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Myocardial Infarction; Diabetes Mellitus, Type 2; Atherosclerosis; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Nordic Diet (Experimental): Dietary advice and provided with some key food items of the healthy Nordic diet
  Interventions: Other: Healthy Nordic Diet
- Usual care (Active Comparator): Dietary advice according to standard clinical care at the cardiology unit
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Other: Healthy Nordic Diet — Participants will be adviced a healthy Nordic diet and will also receive certain Nordic foods high in wholegrains and polyunsaturated fat from vegetable sources
  Arms: Healthy Nordic Diet
Behavioral: Usual Care — Usual care lifestyle advice and national and general recommendations on diet
  Arms: Usual care

SUMMARY:
Diet can play a key role in atherosclerosis and coronary heart disease (CHD), but little interventional data exists, and the mediators of possible anti-atherosclerotic effects of diet are unclear. The investigators will investigate if a healthy Nordic diet (HND) reduces plaque volume, coronary artery calcification (CAC), and plaque inflammation (FAI) in CHD, and examine if changes in gut microbiota may be linked to plaque progression over time. The investigators will also explore if the diet response can be predicted by the metabolic phenotype.

In total 150 CHD patients is randomized to a HND rich in unsaturated fat and fibre from plants, or to a "usual care diet" for 18 months. Plaque volume and composition is assessed by CT, and fecal microbiota composition is determined by deep metagenome shotgun sequencing. CHD and metabolic risk factors, liver fat, muscle fat and biomarkers of diet adherence (plasma fatty acids, whole-grain metabolites) are measured. Machine-learning is used to identify diet "responders" on plaque progression, based on the individual microbiome and metabolome.

If a HND reduces plaque progression, this would be novel information of clinical importance. Also, if the diet alters microbiota that are linked to plaque progression, this would be of high scientific interest. Finally, potential prediction of the diet-response would open up for more personalized treatment of atherosclerosis.

DETAILED DESCRIPTION:
Atherosclerosis of coronary arteries is the main cause of coronary heart disease (CHD). In atherosclerosis, atherogenic lipids are deposited in the arteries to form plaques, and the larger the plaque volume, the more narrowing of the vessel. It is now feasible to directly visualize clinically relevant changes in plaque volume and composition (e.g. calcification, lipid content) by modern computed tomography (CT) angiography. Diet is a cornerstone in both primary and secondary prevention, but it is still not clear if dietary intervention can reduce coronary plaque progression as assessed by modern imaging technique.

In the Nordic countries, a promising alternative to Mediterranean diets is the Healthy Nordic diet. Controlled trials conducted in various Nordic populations have shown that healthy Nordic diets cause reduction of several key CVD risk factors such as elevated blood lipids and blood pressure, hyperglycemia, and inflammation. The Healthy Nordic diet is mainly, but not exclusively, a plant-based diet that accord with the Nordic Nutrition Recommendations (NNR 2023), e.g. is rich in vegetable fats from oils, spreads, nuts and seeds, whole-grains from rye, barley and oats, legumes, vegetables, Nordic fruits and berries but with moderate portions (2-3 times per week) of fatty fish (e.g. Salmon). The effects of a Healthy Nordic diet in a secondary preventive setting and in particular the potential impact on atherosclerosis is yet unknown. The investigators hypothesize that a Healthy Nordic Diet has anti-atherosclerotic properties that can reduce the progress of atherosclerosis and reduce key CVD risk markers and inflammation in patients with a recent MI or chronic coronary syndrome (CCS). Further, the investigators hypothesize this diet will have favorable changes on the gut microbiota, which in turn can contribute to reduced coronary plaque progression.

The overall aim is to compare the ability of a Healthy Nordic Diet versus usual care dietary advice to influence coronary plaque volume and CVD risk after 18 months in patients with MI or with CCS.

The primary aim is to investigate if a Healthy Nordic Diet can reduce plaque volume after 18 months as compared with usual care and routine dietary and lifestyle advice, and secondary aims are to investigate dietary effects on plaque composition, coronary artery calcium (CAC) and coronary inflammation (perivascular fat, fat attenuation index), as well as on ectopic fat content (e.g. liver). Exploratory aims are to investigate the dietary effects on gut microbiota, as well as on metabolomic- lipidomic- and proteomic plasma profiles. In addition, the investigators will monitor blood glucose control using wearable continous glucose monitors (CGMs) as well as Actiheart monitors to record heart ECG and activity with multiple data endpoints.

This study, named NORDHEART, is a randomized, single-blinded, parallel study including a dietary intervention group and a control group, in individuals with diagnosed MI or CCS. The investigators aim to include n=150 individuals in this trial. The majority of participants will be recruited at the Uppsala University hospital but further Swedish recruitment center in mid Sweden might be added if the recruitment rate in Uppsala is slower than expected.

Inclusion criteria include men and women with diagnosed MI from 2 weeks after diagnosis and 6 months after diagnosis, or with CCS (e.g. stable angina pectoris), ages 50 to 80 years, BMI 25-40.

The intervention diet consists of advice to follow a Healthy Nordic Diet as, and it will be advised ad libitum. Certain key food items will be provided (~5 E%) to participants in the intervention. The control group ("usual care") will receive dietary advice in accordance with routine clinical procedures at the cardiology clinic at the Uppsala academic hospital, which follows the national guidelines for lifestyle advice in CVD care.

To monitor dietary intake in both groups, 4-day food records will be conducted at baseline, 6 months, 12 months and 18 months after study entry. Plasma fatty acid composition will be measured to objectively monitor any changes in dietary fat quality, and serum alkylresorcinols will be assessed as valid biomarkers of whole-grain intake from rye and wheat.

The primary outcome is difference between the groups in change in coronary artery plaque volume from baseline to 18 months. Intention-to treat analyses will be the primary analyses.

Secondary outcomes are change in plaque composition and inflammation (perivascular fat and inflammation, coronary calcification [CAC score], liver fat and hepatic fibrosis, LDL-cholesterol, HDL-cholesterol, ApoB, triglycerides, HbA1c, inflammation markers, from baseline to 18months, and a composite of atherosclerotic cardiovascular disease events during the 18 month follow-up.

Exploratory outcomes include effects on gut microbiota, and proteins and lipids (e.g. ceramides) involved in inflammation and markers of the atherosclerotic process. In addition, prediction models using lipidomics, metabolomics, proteomics and genetics will be assessed to explore determinants of responders and non-responders to the dietary intervention, with regard to effects on plaque volume and composition.

The plaque volume and plaque composition with be assessed by novel photon-counting CT angiography (CCTA). This technique can identify and characterize subclinical atherosclerotic disease in most vascular beds, and will be assessed at baseline and 18 months.

Given the large patient group of CHD worldwide, the clinical significance of this study has large potential, especially since there is still only limited evidence to suggest that intense dietary intervention might halt the atherosclerotic progress per se.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Diagnosis with MI from 2 weeks after diagnosis and with maximum 6 months after diagnosis
* Diagnosis with CCS (e.g. stable angina pectoris)
* Ages 50 to 80 years
* BMI 25-40.

Exclusion Criteria:

* Severe heart failure (NYHA classes III, IV)
* Alcohol intake >20g/day
* Unwillingness to follow a new prescribed diet for 18 months
* Other diseases implying a short estimated life expectancy (e.g. severe malignant or kidney or liver disease, as judged by consenting physician).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in coronary plaque volume | 18 months
  Will be assessed by photon-counting CT angiography

SECONDARY OUTCOMES:
Change in coronary inflammation: Fat attenuation Index | 18 months
  Perivascular fat will be assessed by photon counting CT angiography
To investigate if a Healthy Nordic Diet can decrease progression of atherosclerosis Change in coronary artery calcium score (CACS) | 18 months
  CACS will be assessed by photon counting CT angiography
Change in ectopic fat (liver, heart, muscle) | 18 months
  Will be assessed by photon counting CT angiography
Change in blood glycemic control | 6, 12 and 18 months
  Will be measured in fasting state and continously using CGM
Change in plasma LDL cholesterol | 18 months
  Will be assessed by routine methods at the hospital lab
Change in systolic and diastolic blood pressure | 6, 12 and 18 months
Incident cardiovascular events | 18 and 30 months (12 month post intervention)
  A composite outcome will be assesed
Change in hepatic fibrosis | 18 months
  Liver stifness and fibrosis stages assessed by Fibroscan

OTHER OUTCOMES:
Change in gut microbiota | 12 and 18 months
  Gut microbiota will be measured in fecal samples
Change in plasma inflammation proteins | 6, 12 and 18 months
  Protemomic approcah will be used
Change in plasma lipidomic profile including ceramides | 6, 12 and 18 months
  Lipidomic approach will be used
Change in plasma metabolite pattern | 6, 12 and 18months
  A metabolomic approach will be used

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Risérus, MMED, PHD, Principal Investigator — Uppsala University
Locations (1):
- Cardiology clinic, Uppsala university hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided